CLINICAL TRIAL: NCT07392710
Title: Clinical Evaluation of the Nova Max Pro Statsensor Point of Care Creatinine Measuring Device in the Clinical Outpatient and Home Setting & Assessment of the Patient Experience
Brief Title: Clinical Evaluation of the Nova Max Pro StatSensor Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22/NW/0323
Record Dates: First submitted 2026-01-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant; Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The 12-week study involves up to six visits aligned with routine outpatient appointments (about every two weeks). A total of 100 subjects will join the main study, with 30 also participating in a nested sub-study. Subjects are identified during transplant clinic visits and, after written consent, assigned a unique study code accessible only to the research team. As part of standard care, patients have venous blood drawn weekly or fortnightly; the study adds one extra 2ml sample at the same time, totalling up to six samples. At each visit, two capillary samples (finger prick) will be taken using the Nova Max Pro StatSensor device, operated by trained staff, with results recorded in the eCRF. Sub-study participants will use the device at home to measure creatinine within 24 hours of clinic visits (five times), bringing the device to appointments for data retrieval. At the final visit, they will complete a usability survey and a 45-minute interview about their experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study (Other): Assessment of capillary blood creatine levels, using the Nova Max Pro device, at the participating site, on the day of the patient's routine outpatient clinic visit and in the remote setting.
  Interventions: Device: Nova Max Pro StatSensor device

INTERVENTIONS:
Device: Nova Max Pro StatSensor device — The Nova Max Pro StatSensor creatinine analyser is a handheld device used for the quantitative measurement of creatinine in capillary, venous and arterial blood. This study will evaluate the Nova Max Pro in the outpatient setting to ascertain whether the device can be used to reliably monitor renal function remotely post-transplantation.

SUMMARY:
Blood creatinine is an important biomarker used to monitor kidney function. In patients with chronic kidney disease or patients who have received a kidney transplant, careful and frequent monitoring of kidney function is required to enable timely intervention in the event of deteriorating kidney function. Indeed, following kidney transplantation, patients may have their blood serum creatinine checked on average 20 times, during the first year post-transplantation to monitor for graft rejection.

In current clinical practice, most blood creatinine assessments (blood tests) are undertaken in the primary care GP clinics or hospital settings. This practice places burden on healthcare resources and may delay the early detection of deteriorating kidney function. It also places additional burden on patients and impact's their lives as patients are required to attend frequent clinic appointments and undertake regular blood tests. Therefore, the ability for individuals to remotely self-monitor their own kidney function would have a number of health and socio-economic related benefits.

Currently the study will evaluate the clinical usefulness and reliability of a handheld point of care creatinine monitoring device called the Nova Max Pro StatSensor device, in patients who have recently received a kidney transplant. The aim is to compare the clinical performance (i.e accuracy and precision) of the device, with standard laboratory based measurements for measuring blood creatinine levels, in 100 transplant patients attending the outpatient clinic. All patients will be enrolled in the study for a period of 12-weeks. As part of the nested sub-study, 30 participants will measuring their creatinine levels using the Nova Max Pro StatSensor device at home, on the morning of their outpatient clinic. the study will assess the patients experience and attitude towards using the device via a questionnaire and structured interview at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18-year-old
* Able to provide informed consent
* Receipt of a renal transplant
* Attending the renal transplant clinic and the study site.
* Sub-study only: Demonstrate proficiency in using the Nova Max Pro device correctly at Screening (V1) or Visit 3, if enrolling in sub-study at later date.

Exclusion Criteria:

* Declined written informed consent
* Pregnant females or females who plan to conceive during the 12-week study period.
* History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational device, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation (CV) calculated from repeated creatinine measures taken from the Nova Max Pro creatinine analyser and reference laboratory method over the duration of the study | Up to 12 weeks
Mean measurements & standard deviation of repeated creatinine measures taken from the Nova Max Pro creatinine analyser and reference laboratory method over the duration of the study | Up to 12 weeks
A structured questionnaire undertaken at the end of the study will assess subjects' satisfaction and attitudes towards creatinine self-monitoring with the Nova Max Pro creatinine analyser. | Up to 12 weeks
A structured interview undertaken at the end of the study will assess subjects' satisfaction and attitudes towards creatinine self-monitoring with the Nova Max Pro creatinine analyser. | Up to 12 weeks

SECONDARY OUTCOMES:
Coefficient of variation calculated from repeated creatinine measures taken from the Nova Max Pro creatinine analyser and local laboratory over the study period. Results from outpatient and remote settings will be analysed together and separately. | Up to 12 weeks
Mean measurements & standard deviation of repeated creatinine measures taken from the Nova Max Pro device and reference laboratory method over the duration of the study | Up to 12 weeks
Assessed by determining the concordance correlation coefficient for Nova Max Pro creatinine analyser compared with measurements obtained by the laboratory reference methods. Measurements obtained in outpatient and remote settings will be analysed | Up to 12 weeks
R2 and Intraclass correlation coefficient (ICC) for repeated measurements from the Nova Max Pro creatinine analyser. | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Harber, Dr, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD as it will not add any value to publication